CLINICAL TRIAL: NCT06058494
Title: Multi-scale Modeling for Predictive Characterization of Ligaments and Grafts Behavior in ACL Reconstruction
Acronym: MULTI-ACL
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Collaborators: Ministry of Health, Italy (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0023352
Record Dates: First submitted 2016-05-25; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Anterior Cruciate Ligament Reconstruction
Keywords: Anterior Cruciate Ligament; Reconstruction; Ligament modeling
MeSH Terms: interventions — Anterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Single-Bundle: Single-bundle ACL reconstruction
  Interventions: Procedure: Anterior Cruciate Ligament Reconstruction
- Single-Bundle+Lateral Plasty: Single-bundle ACL reconstruction with lateral plasty
  Interventions: Procedure: Anterior Cruciate Ligament Reconstruction
- Double-Bundle: Double-bundle ACL reconstruction
  Interventions: Procedure: Anterior Cruciate Ligament Reconstruction

INTERVENTIONS:
Procedure: Anterior Cruciate Ligament Reconstruction — Reconstruction of the anterior cruciate ligament by means of the three reported techniques, namely single-bundle, single-bundle with extraarticular tenodesis and anatomic double-bundle.

SUMMARY:
The objective of this clinical trial is provide in vivo data thus to model the ligament biomechanical behavior within the physiologically healthy joint and to use the implemented model to predict risk and success rates focusing on knee joint Anterior Cruciate Ligament (ACL) reconstruction. Current ACL surgery offers 3 alternatives: autografts, allografts and bioengineered grafts; the choice of the implant and its characteristics still remains a critical point. The knowledge of patient-specific joint and graft biomechanics is fundamental to reduce surgical revision rate and low functional outcome. This clinical trial will provide data coming from patient-specific biomechanics into a prognostic computational model, able to provide information on both the optimal customized reconstruction and graft status during the early rehabilitation phase. This patient-specific approach will lead to quicker return to sports activity, reducing also the possibility of early osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Primary ACL lesion
* Ability to read and sign the informed consent.
* Age between 16 and 50 years old

Exclusion Criteria:

* Prior surgeries at the same knee
* Grade II or higher lesions at the collateral ligaments
* Posterior Cruciate Ligament lesion
* Inflammatory arthritis or other forms systemic inflammatory diseases
* Local or systemic infections
* Any injury or condition that adversely affects the ability to walk or to participate to I/II level activities
* Previous or concomitant lesions at the contralateral knee
* Skeletal immaturity
* Other potential risk factors for the development of osteoarthritis

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with primary lesion of the anterior cruciate ligament (ACL), assessed by clinical manouvers and confirmed by means of MRI.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Clinical Assessment, Knee Joint Laxity, Kinematics and Dynamics | At baseline
  Active movements will be acquired by dynamic Roentgen Stereophotogrammetric Analysis (RSA) before and after surgery; joint dynamics will be estimated by analyzing Ground Reaction Force, applying inverse dynamics modeling. Navigation system will intra-operatively acquire passive joint kinematics. Clinical assessement will be performed: subjective (KOOS, SF-12) and objective (IKDC, Marx) ones.
Clinical Assessment, Knee Joint Laxity, Kinematics and Dynamics | 4 months
  Active movements will be acquired by dynamic Roentgen Stereophotogrammetric Analysis (RSA) before and after surgery; joint dynamics will be estimated by analyzing Ground Reaction Force, applying inverse dynamics modeling. Navigation system will intra-operatively acquire passive joint kinematics. Clinical assessement will be performed: subjective (KOOS, SF-12) and objective (IKDC, Marx) ones.
Clinical Assessment, Knee Joint Laxity, Kinematics and Dynamics | 18 months
  Active movements will be acquired by dynamic Roentgen Stereophotogrammetric Analysis (RSA) before and after surgery; joint dynamics will be estimated by analyzing Ground Reaction Force, applying inverse dynamics modeling. Navigation system will intra-operatively acquire passive joint kinematics. Clinical assessement will be performed: subjective (KOOS, SF-12) and objective (IKDC, Marx) ones.

SECONDARY OUTCOMES:
Functional and Anatomical Model | at 4 months
  MRI scans with T2 mapping will be performed on each patient to acquire the anatomical features, define the cartilage and graft status.
Functional and Anatomical Model | 18 months
  MRI scans with T2 mapping will be performed on each patient to acquire the anatomical features, define the cartilage and graft status.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Zaffagnini, Prof, MD, Principal Investigator — Istituto Ortopedico Rizzoli; Nicola Francesco Lopomo, Prof, Study Director — Istituto Ortopedico Rizzoli; Cecilia Signorelli, PhD, Study Chair — Istituto Ortopedico Rizzoli; Marco Bontempi, PhD, Study Chair — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Institutional Website — http://www.ior.it